CLINICAL TRIAL: NCT06352203
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Modulating Effect of Probiotics on the Intestinal Microbiota of Pediatric Patients With Neurodevelopmental Disorders.
Brief Title: Effect of Probiotics on the Intestinal Microbiota of Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUT/23.02
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 1 dose of the probiotic every 24 hours, for 6-months.
  Arms: Probiotic
Dietary Supplement: Placebo — 1 dose of the placebo every 24 hours, for 6-months.
  Arms: Placebo

SUMMARY:
Numerous studies have described an altered gut microbiota composition (dysbiosis) in patients with neurodevelopmental disorders that can be correlated with their symptoms, especially gastrointestinal symptoms.

An interventional, randomised, double-blind, placebo-controlled study will be conducted to investigate the effect of a probiotic supplement on the microbiota composition of children aged 3-7 years with neurodevelopmental issues.

The duration of the study will be of 6 months approximately, including 6 months of product intake.

Participants will be randomly assigned to one of the two study groups: control group with placebo administration or probiotic administration group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 7 years old.
* Diagnosed with autism spectrum disorder, according to the clinical criteria of the "Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)" and who meet criteria for ASD according to the ADOS-2 classification.
* Presenting one or more gastrointestinal symptoms (constipation, diarrhoea, abnormal stools, painful defecation, abdominal pain, reflux, bloating, flatulence).
* Written informed consent signed by the parent or legal guardian with express or tacit consent of the other parent.

Exclusion Criteria:

* With intake of antibiotics in the last month.
* With intake of probiotics in the last two weeks.
* Diagnosed with short bowel syndrome or has undergone relevant surgery on the gastrointestinal tract.
* Exhibiting a defect in the intestinal epithelial barrier (e.g. inflammatory bowel disease (IBD)).
* Diagnosed with endocrinological diseases such as diabetes mellitus, hypo- and hyperthyroidism, Cushing's disease, Addison's disease, etc.
* Having heart failure and a cardiac medical history (e.g. artificial heart valve, medical history of infective endocarditis, rheumatic fever, or cardiac malformation).
* Congenital or acquired immunodeficiency.
* Immunocompromised (e.g., cancer and/or transplant patients taking certain immunosuppressive drugs, patients with inherited diseases that affect or may affect the immune system).
* Uncertainty on the part of the investigator about the willingness or ability of the minor's parents or legal guardian to comply with the requirements of the protocol.
* With oral hyper sensitivity impairments that prevent the uptake of the study product.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of children with intestinal dysbiosis after 6 months of treatment. | After 6 months of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infantil Niño Jesús, Madrid, Spain